CLINICAL TRIAL: NCT06284369
Title: Developing, Evaluating and Testing Video Messages for a Smoking Cessation Campaign Among Mongolian Adults
Brief Title: Video Messages for Smoking Cessation Campaign
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This project was determined by LLU IRB to not be human subjects research on 04.10.2024. No subjects were recruited.
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Mongolia
Record Dates: First submitted 2024-02-13; First posted 2024-02-28 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants don't know which video each subject is randomized to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Loss-framed message (Experimental): Loss-framed message. This 54-second video advertisement employs a loss-framed message, highlighting the detrimental costs associated with continued smoking, including the severe negative health impacts such as increased vulnerability to complications from COVID-19 and the likelihood of ICU hospitalization. The main focus of the ad is a well-known young male Mongolian singer, who serves as the central figure conveying the message.
  Interventions: Behavioral: Developing, Evaluating and Testing Video Messages for a Smoking Cessation Campaign
- Gain-framed message (Experimental): Gain-framed message. In this 59-second video advertisement, the emphasis is on highlighting the gains associated with quitting smoking. The narrative follows a female protagonist who, one year after quitting, meets with her physician. The physician highlights the client's improved lung X-ray and blood test results compared to the previous year, offering congratulations on the decision and celebrating the positive health outcome. Encouraged by this progress, the client is motivated to continue making positive lifestyle choices.
  Interventions: Behavioral: Health Message Framing

INTERVENTIONS:
Behavioral: Developing, Evaluating and Testing Video Messages for a Smoking Cessation Campaign — To explore how smokers reacted to the gain-framed and loss-framed video ad
  Other Names: Health message framing effects on attitudes, intentions and behavior
  Arms: Loss-framed message
Behavioral: Health Message Framing — Gain- framed messages in health communication are constructed by framing a particular outcome as either a benefit or a cost, relative to a specific reference poin
  Other Names: Message framing
  Arms: Gain-framed message

SUMMARY:
240 adult smokers will be recruited. Subjects will be asked to view video messages that encourage smoking cessation. The effect of these videos will be assessed.

DETAILED DESCRIPTION:
This study will use a parallel, two-arm randomized control trial design. After consenting to participate in the study, Participants will be invited to fill out the online questionnaire form which will include one randomly selected ad exposure. The participation in the study will contain three parts: pre-test, video-ad stimuli, and post-test. Pretest will contain questions on the demographic information and readiness to quit smoking. Video ad stimuli segment will contain the selected video ad. The posttest will contain the manipulation check, readiness to quit smoking, message engagement, and PME questions. A randomization table will be generated using Research Randomizer software (ResearchRandomizer.org; Social Psychology Network) and subjects will be randomized to video ad 1 or video ad 2 in permuted blocks of 2.

The video ads are a part of the "Victory" media campaign designed for the tobacco cessation clinical project in Mongolia. Each video ad ends with the slogan "Every attempt is a victory".

Video Ad 1. This video ad was designed using a loss-framed message and emphasized the costs of continuing to smoke (losses) demonstrating the severe negative health consequences of smoking (e.g., complicated COVID-19, ICU hospitalization). The main actor in the ad is a famous young male Mongolian singer.

Video Ad 2. The video emphasized the benefits of quitting (gains) using a female actor.

After the viewing of the video ad participants will be asked to report reaction by completing an online posttest survey.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years and older
* Current smoker every day or some days
* Has smoked a minimum of 100 cigarettes in a lifetime

Exclusion Criteria:

* Non Smokers
* Must have internet access to complete questionnaires

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Message Engagement | Immediately post-video message view.
  Subjects will complete a 3 question survey indicating identification with the video message, that will be measured on a 5 point Likert Scale. 1 indicates strong disagreement. 5 indicates strong agreement. The question responses will be added up and a mean will be calculated to create an overall message engagement score.

SECONDARY OUTCOMES:
Readiness to Quit Smoking | Change between pre-exposure and post-exposure to video message, an average of 3 days
  The question will use a 10-point slider to determine how ready a participant is to quit smoking within the next 30 days.

IPD SHARING:
Plan to Share IPD: No